CLINICAL TRIAL: NCT02479971
Title: Effect of Peritoneal Lavage With Clindamycin-gentamicin Solution on Postoperative Pain and Analytic Acute Phase Reactants Following Laparoscopic Sleeve Gastrectomy
Brief Title: Effect of Peritoneal Lavage With Clindamycin-gentamicin on Laparoscopic Sleeve Gastrectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Hospital General Universitario Elche (Other)
Responsible Party: Principal Investigator, Jaime Ruiz-Tovar, MD, PhD, Jaime Ruiz-Tovar, MD, PhD, Hospital General Universitario Elche
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: HGUE 2015-5
Record Dates: First submitted 2015-06-17; First posted 2015-06-24 (Estimated); Last update posted 2015-06-24 (Estimated); Status verified 2015-06

CONDITIONS: Pain
MeSH Terms: conditions — Pain

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Normal saline irrigation (Active Comparator): An irrigation of the entire abdominal cavity with 500 ml normal saline will be performed.
  Interventions: Drug: Normal saline irrigation
- Clindamycin-gentamicin irrigation (Experimental): An irrigation of the entire abdominal cavity with 500 ml gentamicin and clyndamycin solution will be performed.
  Interventions: Drug: Clindamycin-gentamicin irrigation

INTERVENTIONS:
Drug: Clindamycin-gentamicin irrigation — An irrigation of the entire abdominal cavity with 500 ml gentamicin-clindamycin solution will be performed.
  Other Names: Clindamycin-gentamicin solution
  Arms: Clindamycin-gentamicin irrigation
Drug: Normal saline irrigation — An irrigation of the entire abdominal cavity with 500 ml normal saline will be performed.
  Other Names: Saline irrigation
  Arms: Normal saline irrigation

SUMMARY:
A prospective, randomized study will be performed in patients undergoing laparoscopic sleeve gastrectomy (LSG) as bariatric procedure. The patients will be randomized into 2 groups: those patients undergoing an intra-abdominal lavage with normal saline (Group 1) and those undergoing an intra-abdominal lavage with a gentamicin-clindamycin solution (Group 2). Postoperative pain and C reactive protein will be investigated 24 hours after surgery.

DETAILED DESCRIPTION:
A prospective, randomized study will be performedin patients undergoing laparoscopic sleeve gastrectomy (LSG) as bariatric procedure. The patients will be randomized into 2 groups: those patients undergoing an intra-abdominal lavage with normal saline (Group 1) and those undergoing an intra-abdominal lavage with a gentamicin-clindamycin solution (Group 2). Postoperative pain and C reactive protein will be investigated 24 hours after surgery.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) >40 Kg/m2
* BMI > 35 Kg/m2 with the presence of comorbidities associated to obesity
* Patients undergoing laparoscopic sleeve gastrectomy (LSG) as bariatric procedure.

Exclusion Criteria:

* Gastroesophageal reflux
* Preoperative diagnosis of chronic renal failure
* Uncontrolled psychiatric disorders
* Active infections
* Malignancies
* Any other concomitant pathology considered as a contraindication for bariatric surgery.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Postoperative pain | 24 hours after surgery
  Postoperative pain will be evaluated by a Visual Analogic Scale 24 hours after surgery

SECONDARY OUTCOMES:
C reactive protein | 24 hours after surgery
  C reactive protein will be evaluated at a blood analoytics obtained 24 hours after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Arroyo, MD, PhD, Study Director — Hospital general Elche